CLINICAL TRIAL: NCT01496508
Title: Principal Investigator
Brief Title: High-frequency Oscillatory Ventilation (HFOV) in Preterm Infants With Severe Respiratory Distress Syndrome (RDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhengzhou Children's Hospital, China (Other)
Responsible Party: Principal Investigator, Changlian Zhu, Professor, Zhengzhou Children's Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZZ-HFOV
Record Dates: First submitted 2011-12-13; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: high-frequency oscillatory ventilation; respiratory distress syndrome; preterm infants; neurodevelopment; preterm infants with severe respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFOV (Experimental): A SLE5000 infant ventilator was used as the high-frequency ventilator.HFOV setting were as follows: initial frequency was set between 11 and 15Hz; pressure amplitude of oscillation was initially adjusted to provide adequate chest wall movement and was subsequently titrated to maintain the PaCO2 between 40 and 55 mmHg.Extubation was considered when the patient's condition was stable for 12-24h, while adequate oxygenation could be maintained with an FIO2 <0.3 and respiratory rate <25/min.
  Interventions: Device: mechanical ventilation (SLE 5000, Servo-i-Maquet)
- CV (Experimental): A Servo-i-Maquet will be used as the conventional mechanical ventilator. CV settings were: exhaled tidal volumes set at 5-6 mL/kg, initial peak inspiratory pressure (PIP) of 15-25 cmH2O; positive expiratory end pressure (PEEP) set to 4-6 cmH2O; inspiratory times of 0.25-0.40s; rates set to <60/min. The weaning process was initiated when the following parameters were achieved: PIP <18 cmH2O, PEEP <4 cmH2O, and FIO2 <0.4. Extubation was considered when the patient's condition was stable for 12-24h, while adequate oxygenation could be maintained with an FIO2 <0.3 and respiratory rate <25/min. All infants extubated onto nasal continuous positive airway pressure (Infant Flow, Electro Medical Equipment) and then weaned to a nasal cannula, and then to room air.
  Interventions: Device: mechanical ventilation (SLE 5000, Servo-i-Maquet)

INTERVENTIONS:
Device: mechanical ventilation (SLE 5000, Servo-i-Maquet) — Ventilation strategies for both groups were to emphasize lung recruitment and avoid atelectasis and over distention. The optimum lung volume was determined as expansion to 8 to 9.5 ribs for most infants, and 7 to 8 ribs for infants with air leak. HFOV setting were as follows: initial frequency was set between 11 and 15Hz; pressure amplitude of oscillation was initially adjusted to provide adequate chest wall movement and was subsequently titrated to maintain the PaCO2 between 40 and 55 mmHg; The initial mean airway pressure (MAP) was set at 8-10 cmH2O. MAP and FIO2 were set to maintain arterial oxygen saturation between 88 to 95%, an arterial pH of at least 7.25. Extubation was considered when MAP was ≤7 cmH2O and the pressure amplitude of oscillation reach 10 to 15 cmH2O.
  Other Names: conventional mechanical ventilation

SUMMARY:
Respiratory distress syndrome (RDS) is common in preterm infants born at less than 32 weeks gestation; surfactant and mechanical ventilation have been the standard treatment. However, despite advances in neonatal respiratory care, a considerable number of preterm infants develop chronic lung disease, termed bronchopulmonary dysplasia (BPD), which is associated with neonatal death, prolonged neonatal intensive care stay, and impaired neurodevelopment. High-frequency oscillatory ventilation (HFOV) was developed as a new ventilation technique in the late 1970s. It was expected to result in less BPD and death as a primary model of ventilation compared to conventional ventilation (CV) in the treatment of RDS. However, there is disagreement concerning the advantage of HFOV over CV in the treatment of RDS in preterm infants regarding the prevention of death, BPD, intraventricular hemorrhage, and periventricular leucomalacia in the short term. The purpose of this study was to compare the efficacy and safety of HFOV and CV in preterm infants with severe RDS.

DETAILED DESCRIPTION:
All patients were monitored including blood pressure, heart rate, oxygen saturation, ventilator settings, and arterial blood gases pre- or during mechanical ventilation. PaO2/FIO2 was calculated. After 2 hours ventilation, if PaO2/FIO2 <200, patients were given rescue surfactant therapy (Curosurf 200mg/kg). A subsequent dose (100mg/kg) was administered when PaO2/FIO2 <200 12 hours after the previous dose. Surfactant was administered with use of in-line catheters. Suctioning was performed 6 hours after surfactant administration, except for some patients needed suction soon, with use of an in-line suction catheter. Ventilation continued during the administration of surfactant and suctioning.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants admitted to the NICU with gestational age <32 weeks, birth weight <1500g and less than 24 hours of age
2. Who developed RDS requiring mechanical ventilation
3. Presented a partial pressure of oxygen (PaO2): fraction of inspired oxygen (FIO2) ratio <200
4. Radiograph criteria of severe RDS

Exclusion Criteria:

1. Infants with genetic metabolic diseases
2. Congenital abnormalities
3. Pneumothorax
4. Grade III-IV intracranial hemorrhage

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of bronchopulmonary dysplasia | defined as requirement of oxygen at 36 weeks of postmenstrual age
  To count the number of patients with bronchopulmonary dysplasia at 36 weeks of postmenstrual age.

SECONDARY OUTCOMES:
duration of mechanical ventilation | number of days on mechanical ventilation after birth to 36weeks of postmenstrual age
  To calculate how many days of the newborn baby with mechanical ventilation either HFOV or CV at 36 weeks postmenstrual age.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xiong, MD, Study Director — Zhengzhou Children's Hospital
Locations (1):
- Zhengzhou Children's Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Sun H, Cheng R, Kang W, Xiong H, Zhou C, Zhang Y, Wang X, Zhu C. High-frequency oscillatory ventilation versus synchronized intermittent mandatory ventilation plus pressure support in preterm infants with severe respiratory distress syndrome. Respir Care. 2014 Feb;59(2):159-69. doi: 10.4187/respcare.02382. Epub 2013 Jun 13. PMID 23764865